CLINICAL TRIAL: NCT05619016
Title: Phase II Study of [68Ga]Ga-ABY-025 PET for Non-invasive Quantification of HER2-status in Solid Tumors
Brief Title: [68Ga]Ga-ABY-025 PET for Quantification of HER2-status in Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Rimma Axelsson, Professor, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K 2020-9716; 2022-500448-39-00 (Other: EU CT Number)
Record Dates: First submitted 2022-11-07; First posted 2022-11-16 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Neoplasms; Gastric Neoplasms Malignant; Breast Cancer; HER2-positive Gastric Cancer
Keywords: 68-Ga ABY-025; HER2 PET; PET/CT; Gastroesophageal cancer; Metastatic breast cancer; HER2 low
MeSH Terms: conditions — Esophageal Neoplasms; Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-blinded, diagnostic explorative phase II basket trial.
  Investigators select subjects that are scheduled for anti-HER2 treatment due to
  * metastatic HER2 positive gastroesophageal cancer (GEAC)
  * metastatic breast cancer with low HER2 expression (HER2low mBC).
  All patients undergo a PET/CT with the interventional drug/radiotracer 68Ga-ABY-025 before starting treatment. GEAC patients will undergo an additional ABY-025-PET after 3 cycles of treatment. Results will be compared to HER2 analysis of tissue samples.
Masking Description: Treating clinicians will be blinded for the results of the HER2-PET
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with HER2 positive GEAC or HER2 low cancer (pilot) (Experimental): The participants of the study will undergo two sessions of HER2 PET and one 18F-FDG PET/CT for study purposes. The first HER2 PET is performed within 21 days before initiation of the systemic oncological treatment including HER2-targeted drugs, and is followed by tumor biopsies. A second HER2 PET and a second 18F-FDG PET will be performed adjacent to response evaluation after 3 courses of oncological therapy. Data from the PET investigations will be compared to HER2 expression analyses of the biopsy specimen and correlated to disease and survival data at follow up one year after inclusion.
  Within the pilot study, participants with HER2 low mBC will undergo one HER2 PET followed by biopsies.
  Interventions: Diagnostic Test: [68Ga]Ga-ABY-025 PET; Diagnostic Test: Biopsy and analysis of HER2 expression

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-ABY-025 PET — [68Ga]Ga-ABY-025 PET: Each patient in Cohort 1 will be imaged with a PET/CT twice using the radiolabeled investigational product ABY-025 as a tracer. At the time of injection, a 45-minutes long dynamic scan will take place over a pre specified region of interest. Three hours after injection a full body PET scan followed by a CT scan will be performed.
  Other Names: HER2 PET
Diagnostic Test: Biopsy and analysis of HER2 expression — Biopsy: Within 3 days after the first ABY-025-PET a tissue sample from at least one metastasis >10 mm available for biopsy, preferably shallow lymph nodes, will be analyzed for HER2 expression through immunohistochemistry- (IHC) and in situ hybridization- (ISH) analysis in patients with GEAC and HER2low mBC.

SUMMARY:
The goal of this phase II clinical trial is to improve the selection of patients with solid tumors who would benefit from effective treatment with HER2 targeted drugs. This will be achieved by examining patients with HER2 positive tumors in the esophagus or stomach or patients with advanced breast cancer with low HER2 expression (HER2low) with the HER2 specific positron emission tomography (PET) tracer ABY-025 (HER2-PET) and compare the imaging results with HER2 expression in tumor tissue derived from biopsies (reference standard).

DETAILED DESCRIPTION:
The goal of this phase II interventional clinical trial is to evaluate the HER2-status in tumor lesions measured by Gallium-68-ABY-025-uptake on PET/CT with HER2-status defined by reference standard (laboratory analyses) in patients with gastroesophageal cancer (GEAC) and metastatic breast cancer with low HER2 expression (HER2-low mBC).

The participants in GEAC cohort of the study will undergo two sessions of HER2 PET and one 18-Fluorodeoxyglucose (18F-FDG) PET/CT for study purposes. The first HER2 PET is performed within 21 days before initiation of the systemic oncological treatment and is followed by tumor biopsies. A second HER2 PET and a second 18F-FDG PET will be performed adjacent to response evaluation after 3 courses of oncological therapy. Data from the PET investigations will be compared to HER2 expression analyses of the biopsy specimen and correlated to disease and survival data at follow up one year after inclusion. Within the pilot study, participants with HER2 low mBC will undergo one HER2 PET followed by biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. The subject has given written consent to participate in the study.
3. Patients with metastatic disease because of gastroesophageal adenocarcinoma or HER2-low breast cancer. Cohort 1: Histologically confirmed HER2-positive primary gastroesophageal adenocarcinoma, scheduled for palliative HER2-targeted therapy; Cohort 2: HER2-low metastatic breast cancer first within a pilot study (of which five patients with de novo HER2-low mBC and five patients with pre-treated HER2-low mBC). Later, within a post-pilot study. Definition of HER2 positivity (ASCO College of American Pathologist 2018. HER2 Testing for Breast Cancer Guidelines.) HER2-low mBC is defined as IHC 1+ or IHC 2+ but ISH negative.
4. At least one metastatic lesion ≥ 10 mm is available for biopsy defined on CT.
5. At least one (and up to five) additional metastatic index lesion/s ≥ 10 mm for evaluation of treatment effect
6. World Health Organization (WHO) performance status ≤ 2.
7. Expected survival > 12 weeks.

Exclusion Criteria:

1. Significantly impaired renal function (GFR <30 ml/min/1.73 m2)
2. Allergy to iodinated contrast media
3. Subjects that for some reason are unable to exercise their rights, such as cognitive function impairment.
4. Other manifest malignancy except for basal cell carcinoma of the skin.
5. The patient presenting any contraindication for the use of HER2 targeted therapy for metastatic disease: congestive heart failure, baseline left ventricular ejection fraction (LVEF) less than 50%, transmural myocardial infarction, uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg), angina pectoris requiring medication, clinically significant valvular heart disease, high-risk arrhythmias, lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome, active gastrointestinal bleeding.
6. Inadequate organ function, suggested by the following laboratory results: absolute neutrophil count <1,500 cells/mm3, haemoglobin <90 g/L, total bilirubin ≥1.5 x Upper Limit of Normal (ULN) (unless the patient has documented Gilbert's syndrome), Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or Alanine aminotransferase (ALT)/ serum glutamic pyruvic transaminase (SGPT) >5.0 x ULN.
7. Positive pregnancy test in women of childbearing potential (premenopausal or <12 months of amenorrhea post-menopause and who have not undergone surgical sterilization), or lactation.
8. Female patients of childbearing potential and sexually active and not willing to use a highly effective contraceptive. Examples of highly effective contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone releasing intrauterine devices (IUDs), and copper IUDs. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. Women must refrain from donating eggs during this same period.
9. Patients with increased risk of complications from biopsies, i.e. increased risk of bleeding, defined as

   * prothrombin time test (INR value) >1.4, platelet count <70 (109/l), activated partial thromboplastin time (APTT) >30s.
   * known bleeding disorder such as hemophilia, von Willebrand disease or platelet disorders.
   * any anticoagulants or antiplatelet treatment (except for low-dose acetyl-salicylic acid (ASA), i. e 75 mg daily).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of HER2-positive lesions | up to 24 months
  Percentage of HER2-positive lesions (primary tumors and/or metastases) measured by tracer uptake on PET/CT which are also positive regarding HER2-status defined by reference biopsy-based standard used in clinical routine in patients with GEAC

SECONDARY OUTCOMES:
SUV | up to 24 months
  Optimal Standardized Uptake Values (SUVs) cut-off values for separating HER2-positive/or HER2-low from HER2-negative lesions by reference standard methods.
TBR | up to 24 months
  Tumor-to-Background Ratio (TBR) cut-off values for separating HER2-positive/or HER2-low from HER2-negative lesions by reference standard methods.
Intra-individual heterogeneity of HER2-positivity | up to 24 months
  Percentage of tracer uptake sites on whole-body HER2 PET compared to all known cancer-related lesions, determined on the routine radiological investigation with CT as an estimation of intra-individual heterogeneity of HER2-positivity.
Feasibility in HER2low | up to 24 months
  Percentage of false-negative findings on HER2 PET compared to results from immunohistochemistry testing (IHC) from at least one index lesion in patients with HER2-low mBC.
HER2 positive cancer burden | up to 24 months
  Percentage of tracer uptake in sites, not previously determined on the routine radiological investigation with CT, as a measure of cancer burden determined on the whole body HER2 PET in tumor lesions.
Safety aspects of ABY-025 | up to 36 months
  Frequency of Adverse Events (AEs), Adverse Reactions (ARs), Serious Adverse Events (SAEs), and Suspected Unexpected Serious Adverse Reactions (SUSARs).

OTHER OUTCOMES:
Treatment response 1 | up to 36 months
  To examine the change in HER2 expression measured by tracer uptake on PET/CT (SUVs and TBR) performed after 3 courses of chemotherapy/HER2 targeted drugs compared to pre-treatment values and in which proportion of the examined patients this occur.
Treatment response 2 | up to 36 months
  Changes in SUVs in index lesions, as well as in the total HER2-positive tumor volume at HER2 PET (percentage) before and after treatment with systemic therapy including HER2 targeted drugs to evaluate treatment response.
Comparison between HER2 PET and FDG PET | up to 24 months
  Comparison of treatment response evaluation performed by HER2 PET versus 18F-FDG PET/CT defined as percentage of complete and partial response, stable and progressive disease (percentage of concordant results).
HER2 PET as a prognostic tool | up to 36 months
  The correlation between HER2 expression measured by a total HER2-positive tumor volume at HER2 PET before treatment and progression-free survival (PFS), overall (or clinical) response rate to systemic therapy (ORR) at 12 months after inclusion.
HER2 PET as a marker for treatment related cardiotoxicity | up to 36 months
  The presence and frequency of myocardial uptake of [68Ga]Ga-ABY-025 and relation to treatment-related cardiotoxicity determined by echocardiography.
Dynamic PET parameters | up to 36 months
  The agreement between whole body static imaging and kinetic parameters in the determination of HER2-status.

CONTACTS AND LOCATIONS:
Overall Officials: Rimma Axelsson, Prof., MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Department of Radiation Physics and Nuclear Medicine, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Velikyan I, Schweighofer P, Feldwisch J, Seemann J, Frejd FY, Lindman H, Sorensen J. Diagnostic HER2-binding radiopharmaceutical, [68Ga]Ga-ABY-025, for routine clinical use in breast cancer patients. Am J Nucl Med Mol Imaging. 2019 Feb 15;9(1):12-23. eCollection 2019. PMID 30911434
- [Background] Alhuseinalkhudhur A, Lubberink M, Lindman H, Tolmachev V, Frejd FY, Feldwisch J, Velikyan I, Sorensen J. Kinetic analysis of HER2-binding ABY-025 Affibody molecule using dynamic PET in patients with metastatic breast cancer. EJNMMI Res. 2020 Mar 23;10(1):21. doi: 10.1186/s13550-020-0603-9. PMID 32201920
- [Background] Ahlgren S, Orlova A, Wallberg H, Hansson M, Sandstrom M, Lewsley R, Wennborg A, Abrahmsen L, Tolmachev V, Feldwisch J. Targeting of HER2-expressing tumors using 111In-ABY-025, a second-generation affibody molecule with a fundamentally reengineered scaffold. J Nucl Med. 2010 Jul;51(7):1131-8. doi: 10.2967/jnumed.109.073346. Epub 2010 Jun 16. PMID 20554729
- [Background] Sandstrom M, Lindskog K, Velikyan I, Wennborg A, Feldwisch J, Sandberg D, Tolmachev V, Orlova A, Sorensen J, Carlsson J, Lindman H, Lubberink M. Biodistribution and Radiation Dosimetry of the Anti-HER2 Affibody Molecule 68Ga-ABY-025 in Breast Cancer Patients. J Nucl Med. 2016 Jun;57(6):867-71. doi: 10.2967/jnumed.115.169342. Epub 2016 Feb 9. PMID 26912439
- [Background] Sorensen J, Sandberg D, Sandstrom M, Wennborg A, Feldwisch J, Tolmachev V, Astrom G, Lubberink M, Garske-Roman U, Carlsson J, Lindman H. First-in-human molecular imaging of HER2 expression in breast cancer metastases using the 111In-ABY-025 affibody molecule. J Nucl Med. 2014 May;55(5):730-5. doi: 10.2967/jnumed.113.131243. Epub 2014 Mar 24. PMID 24665085
- [Background] Sorensen J, Velikyan I, Sandberg D, Wennborg A, Feldwisch J, Tolmachev V, Orlova A, Sandstrom M, Lubberink M, Olofsson H, Carlsson J, Lindman H. Measuring HER2-Receptor Expression In Metastatic Breast Cancer Using [68Ga]ABY-025 Affibody PET/CT. Theranostics. 2016 Jan 1;6(2):262-71. doi: 10.7150/thno.13502. eCollection 2016. PMID 26877784
- [Background] Tolmachev V, Velikyan I, Sandstrom M, Orlova A. A HER2-binding Affibody molecule labelled with 68Ga for PET imaging: direct in vivo comparison with the 111In-labelled analogue. Eur J Nucl Med Mol Imaging. 2010 Jul;37(7):1356-67. doi: 10.1007/s00259-009-1367-7. Epub 2010 Feb 4. PMID 20130858
- [Background] Sandberg D, Tolmachev V, Velikyan I, Olofsson H, Wennborg A, Feldwisch J, Carlsson J, Lindman H, Sorensen J. Intra-image referencing for simplified assessment of HER2-expression in breast cancer metastases using the Affibody molecule ABY-025 with PET and SPECT. Eur J Nucl Med Mol Imaging. 2017 Aug;44(8):1337-1346. doi: 10.1007/s00259-017-3650-3. Epub 2017 Mar 6. PMID 28261749
- [Derived] Jussing E, Ferrat M, Moein MM, Alfredeen H, Tegnebratt T, Bratteby K, Samen E, Feldwisch J, Altena R, Axelsson R, Tran TA. Optimized, automated and cGMP-compliant synthesis of the HER2 targeting [68Ga]Ga-ABY-025 tracer. EJNMMI Radiopharm Chem. 2023 Nov 22;8(1):41. doi: 10.1186/s41181-023-00226-y. PMID 37991639